CLINICAL TRIAL: NCT06805474
Title: A Prospective Observational Study to Assess the Reliability and Validity of the Multi-Luminance Shape Discrimination Test (MLSDT) With 9 Objects
Brief Title: A Prospective Observational Study to Assess the Reliability and Validity of the MLSDT
Status: Recruiting | Type: Observational
Sponsor: Nanoscope Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NTXOBS-002
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Macular Degeneration; Geographic Atrophy; Stargardt Disease
Keywords: Multi-Luminance Shape Discrimination Test; low-vision magnifying aid (eGlasses); best-corrected visual acuity (BCVA); Early Treatment Diabetic Retinopathy Study ETDRS
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy; Stargardt Disease | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1:: Normal-Sighted Participants with clinically normal ocular findings and BCVA range 20/16 to <20/40 (ETDRS letter score 71 - 90) in each eye.
  Interventions: Other: Observational
- Cohort 2: Moderately Sight-Impaired Participants with a BCVA range of 20/40 to <20/200 (ETDRS letter score of 36 - 70) and a clinical diagnosis of STGD/GA.
  Interventions: Other: Observational
- Cohort 3: Severely Sight-Impaired Participants with a BCVA range of 20/200 to 20/800 (ETDRS letter score of 5 - 35) and a clinical diagnosis of advanced STGD/GA.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The goal of this observational study is to assess the reliability and validity of the 9-object MLSDT for evaluation of participants with moderate to severe vision impairment when tested without a wearable low-vision magnifying aid (eGlasses) and then with eGlasses. These results will be compared to ETDRS testing results for the same participants without eGlasses and then with eGlasses. Two cohorts will consist of participants who have vision loss due to STGD or geographic atrophy (GA) due to age-related macular degenerations (AMD). Normally sighted participants will provide a control group.

DETAILED DESCRIPTION:
Here, we aim to test the accuracy and validate the MLSDT using 9 shapes (instead of 3 shapes) as a reliable, standardized and efficient test of functional vision in STGD and GA patients with impaired vision. This includes evaluation of the performance (retest variability and repeatability) of the test(s) based on patients' visual acuity. Furthermore, we will explore descriptive relationships between MLSDT with best-corrected visual acuity (BCVA) using the Early Treatment Diabetic Retinopathy Study ETDRS) eye chart.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age ≥ 18 years
* Able to comprehend and give informed consent.
* Able to comply with testing and all protocol tests.
* Eligible for 1 of 3 cohorts listed below:

Cohort 1: Normal-Sighted Participants with clinically normal ocular findings and BCVA range 20/16 to <20/40 in each eye (ETDRS letter score 71 - 90) Cohort 2: Moderately-Sight Impaired Participants with a BCVA range of 20/40 to <20/200 (ETDRS letter score of 36 - 70) and a clinical diagnosis of STGD/GA Cohort 3: Severely-Sight Impaired Participants with a BCVA range of 20/200 to 20/800 (ETDRS letter score of 5 - 35) and a clinical diagnosis of advanced STGD/GA

* Clinical diagnosis of STGD for cohorts 2 and 3
* Clinical diagnosis for GA (due to AMD) for cohorts 2 and 3
* Participants who have had anti-VEGF therapy 2 weeks prior to enrollment have to demonstrate 3 months of vision stability and be fluid free on OCT.

Exclusion Criteria:

* Concurrent participation in any interventional clinical trial or receipt of an investigational drug within the previous 6 months

  * Presence of any condition other than STGD or GA from AMD on slit lamp exam or dilated ophthalmoscopy that impairs visual acuity or visual fields e.g., corneal opacity, visually significant cataract or visual field loss in glaucoma
  * No intra-vitreal injection with anti-VEGF two weeks prior to the study
  * Presence of neurological condition that impairs visual acuity
  * Individuals who refuse or are incapable of performing the MLSDT of BCVA tests
  * Individuals with retinal prosthesis (such as ARGUS-II)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll approximately 30 adult participants, to one of 3 cohorts. Participants who meet all the inclusion criteria and for whom none of the exclusion criteria apply will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-27 (Estimated)

PRIMARY OUTCOMES:
MLSDT scores in normal and severely visually impaired subjects with a clinical diagnosis of Stargardt Disease or Geographic Atrophy on MLSDT | 15 days
  Comparison of vision test scores against the ETDRS visual acuity test

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Barone, MD, Study Chair — Nanoscope Therapeutics Inc.
Locations (1):
- Retina of North Texas,, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
The results of the clinical trial will be made available when the study is completed. The results will be published on this site and be available to conference presentations and publications.